CLINICAL TRIAL: NCT02719873
Title: The Impact of Maternal Obesity on Pregnancy Outcomes in El-Minia Locality a Case Control Survey Study
Brief Title: The Impact of Maternal Obesity on Pregnancy Outcomes in El-Minia Locality
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Reham Elkhateeb, doctor, Minia University
Other Study IDs: MOI in pregnancy outcome
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Obesity During Pregnancy in Clinical Practice
Keywords: obesity , pregnancy , maternal and fetal outcome
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control group: the group with normal BMI
- study group: The group with the BMI more than 24.9 kg per meter square to study the impact of maternal obesity in pregnancy outcome
  Interventions: Other: The impact of maternal obesity on pregnancy outcomes

INTERVENTIONS:
Other: The impact of maternal obesity on pregnancy outcomes — observation of maternal obesity effect in foetal and maternal outcome
  Groups: study group

SUMMARY:
A study will carried out over a period of one year , all obese pregnant women as diagnosed with BMI at the time of 1st ANC visit and before labor ,observation of events during both intra-partum &postpartum periods it will be recorded.outcome will compared with normal other pregnant women

DETAILED DESCRIPTION:
It is known that obesity during pregnancy has drawbacks for both maternal and foetal outcome The aim of this study is to evaluate and measure the proportion of the adverse pregnancy outcomes attributable to maternal obesity and so reaching to recommendations in order to improve the outcomes and wellbeing of these women and their children.patient will be divided into two groups control group with normal BMI and study group and both compared as regard foetal and maternal outcome The assessed fetal variables will be: fetal birthweight & incubators admission. Data will be retrieved from patients before labor and from investigator observation both intrapartum and postpartum.

ELIGIBILITY:
Inclusion Criteria:

* obese
* pregnant
* age 18 -40
* single viable cephalic foetus

Exclusion Criteria:

less than 18 years more than 40 years associated medical disorders patient refusal non cephalic presentation

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women with BMI more than 24 per meter square body surface area
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Mode of delivery | onset of labor till end
  vaginal or Cesarean section
shoulder dystocia | 1 minute after delivery of the head
  arrest of shoulder more than one minute after delivery of the head
foetal macrosomia | at time of labour or elective CS
  foetal weight at time of delivery more than 90th percentil

SECONDARY OUTCOMES:
postpartum hemorrhage | onset of labor and for 6 weeks after
  primary or secondary blood loss through birth canal more than 500cc
postpatum maternal infection | end of labor and for 6weeks after
  postpartum signs of sepsis
neonatal ICU admission | one month after delivery
  neonatal ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stuber TN, Kunzel EC, Zollner U, Rehn M, Wockel A, Honig A. Prevalence and Associated Risk Factors for Obesity During Pregnancy Over Time. Geburtshilfe Frauenheilkd. 2015 Sep;75(9):923-928. doi: 10.1055/s-0035-1557868. PMID 26500368